CLINICAL TRIAL: NCT02539147
Title: Characterization of Non-canonical Way in Inflammasome Monocytes of Patients With Severe Sepsis
Acronym: CASPASEs
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Institut Pasteur (Industry); Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A01617-38
Record Dates: First submitted 2015-08-21; First posted 2015-09-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2015-08

CONDITIONS: Severe Sepsis
Keywords: lipopolysaccharide; sepsis; caspase-4 and -5; monocytes; IL-1β and IL-1α
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: None Retained — arterial blood (20ml)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with severe sepsis: blood samples from patients with severe sepsis
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — Isolation and stimulation of monocytes, preparation of cell lysates, measurement of cytokine production, Western blot

SUMMARY:
Activation of caspase-4 and human caspase-5 (orthologs of caspase-11 in mice) in innate immune cells.

DETAILED DESCRIPTION:
Lipopolysaccharide (LPS) of the wall of Gram-negative bacteria is one of pathogen associated molecular patterns (PAMPs), which are recognized by cells of the innate immune system via Toll-like receptor 4 (TLR4) . The LPS / TLR4 interaction induces the secretion of a variety of proinflammatory cytokines. Among them, interleukin-1β (IL-1β) is a major cytokine, and alterations to its secretion has been associated with various diseases, such as periodic syndrome associated cryopyrin (CAPS), gout, rheumatoid arthritis or multiple sclerosis.

The release of IL-1β is controlled by a molecular platform protein, known as the inflammasome name. The canonical protein (that is to say conserved in evolution) of the inflammasome NLRP3 are NLRC4 and that engages the ASC adapter protein to activate caspase-1, which promotes the cleavage of interleukin IL-1β. Gram-negative bacteria such as Escherichia coli cause non-canonical activation of caspase-1, caspase-11In involving more NLRP3 and AUC. In mouse, caspase-11 is essential to the immune response to gram-negative bacteria, but bacterial PAMPs that are responsible for triggering of the non-canonical inflammasome remain to be identified. It has recently been shown that caspase-11 is involved in the death of the mice subjected to septic shock. The mouse model requires caspase-11-dependent mechanism, caspase-independent -1 since the CASP1 - / - mouses are also susceptible to LPS as wild type mice. A key question to be answered is whether LPS triggers similar events in human cells. If this is the case, this knowledge may be useful in drug development for treatment of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* patients with sepsis severe (bacterial infection associated with deterioration of at least one vital function) defined according to the criteria consensus conference
* patients whose diagnosis is made within 24 hours of the opening hours of Pasteur Research Laboratory
* patients with arterial catheter (not to impose an additional puncture to the patient) will be recruited in the intensive care unit of the Hospital St. Joseph. Arterial blood (20 ml) will be charged within 24 hours of the onset of severe sepsis criteria, during working hours of the laboratory of the Pasteur Institute, using vacuum tubes under heparin (Vacutainer), sent by a courier within 2 hours following the removal (to ensure that the cells are sufficiently "fresh" during processing in the laboratory)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sepsis severe (bacterial infection associated with deterioration of at least one vital function) defined according to the criteria consensus conference
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Characterize the expression of caspase-4 and -5 in by measuring the production of cytokines: IL-1β concentrations and IL-1α will determined by ELISA in the cell supernatant will be collected from monocytes stimulated or not | Two hours after blood collection : isolation and stimulation of monocytes than preparation of cell lysates

SECONDARY OUTCOMES:
Correlate the activation of caspases-4 and -5 with IL-1β production with (canonical inflammasome) and IL-1α (Non-canonical inflammasome) measured by Western blot | Two hours after blood collection : isolation and stimulation of monocytes than preparation of cell lysates

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Misset, Professor, Principal Investigator — Fondation Hôpital Saint-Joseph; Jean Marc Cavaillon, Professor, Principal Investigator — Unité Cytokines et Inflammation, Institut Pasteur, Paris; Alessandra Mortellaro, Principal Investigator — Singapore Immunology Network, Agency for Science, Technology and Research, 8A Biomedical Grove, #04-06 Immunos, Singapore
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

REFERENCES:
- [Background] Conforti-Andreoni C, Ricciardi-Castagnoli P, Mortellaro A. The inflammasomes in health and disease: from genetics to molecular mechanisms of autoinflammation and beyond. Cell Mol Immunol. 2011 Mar;8(2):135-45. doi: 10.1038/cmi.2010.81. Epub 2011 Jan 24. PMID 21258359
- [Background] Zambetti LP, Laudisi F, Licandro G, Ricciardi-Castagnoli P, Mortellaro A. The rhapsody of NLRPs: master players of inflammation...and a lot more. Immunol Res. 2012 Sep;53(1-3):78-90. doi: 10.1007/s12026-012-8272-z. PMID 22427013
- [Background] Vigano E, Mortellaro A. Caspase-11: the driving factor for noncanonical inflammasomes. Eur J Immunol. 2013 Sep;43(9):2240-5. doi: 10.1002/eji.201343800. PMID 24037676
- [Background] Kayagaki N, Warming S, Lamkanfi M, Vande Walle L, Louie S, Dong J, Newton K, Qu Y, Liu J, Heldens S, Zhang J, Lee WP, Roose-Girma M, Dixit VM. Non-canonical inflammasome activation targets caspase-11. Nature. 2011 Oct 16;479(7371):117-21. doi: 10.1038/nature10558. PMID 22002608
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622